CLINICAL TRIAL: NCT00224380
Title: Medication Adherence in Older Adults
Brief Title: Medication Adherence in Older Adults With Serious Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Janssen, LP (Industry); National Alliance for Research on Schizophrenia and Depression (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: MA200316456
Record Dates: First submitted 2005-09-15; First posted 2005-09-23 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Schizophrenia; Bipolar Disorder; Depression
Keywords: Serious mental illness; medication adherence
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Depression; Medication Adherence

INTERVENTIONS:
Behavioral: Using Medications Effectively

SUMMARY:
The goal of this pilot study is to learn about how well older people with serious mental illness (including schizophrenia, schizoaffective disorder, bipolar disorder, major depression) follow prescribed medication regimens, and to evaluate a manualized intervention designed to enhance medication management skills and adherence, the Using Medications Effectively program. The following four hypotheses will be tested:

1. Medication adherence will be associated with several variables including insight, memory, medication management skill, knowledge about medications, attitudes about medications.
2. People who receive the program will have better medication adherence compared to those who do not receive the program as measured by pill counts.
3. People who receive the program will develop better medication management skills compared to those who do not receive the program.

DETAILED DESCRIPTION:
Individuals who are already participating in a study of a combined skills training and health care management intervention for older people with serious mental illness are invited to join this study. Half of the individuals have already been randomly assigned to receive the intervention and half have already been randomly assigned to continue receiving their usual care. The people receiving the intervention receive the skills training module, Using Medications Effectively, in 8 group sessions over 8 weeks. The module includes information about common medications used for psychiatric and medical illnesses; training on using devices to help take medications properly; and instruction on strategies to help incorporate medication taking into a daily routine. A trained research assistant conducts pill counts and interview sessions with all participants after they sign an informed consent form, 8 weeks later, and 3 months after the second interview.

ELIGIBILITY:
Inclusion Criteria:

Participation in Rehabilitation and Health Care for Older People with SMI Serious mental illness (schizophrenia, schizoaffective disorder, bipolar disorder, major depression) and functional impairment Receiving mental health services for 3 months or more Age 50 or older Ability to provide informed consent or guardian consent -

Exclusion Criteria:

Currently residing in an institution Psychiatric illness caused by co-morbid medical condition Dementia or score<20 on Mini Mental State Exam

-

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72
Dates: Start 2003-07; Study Completion 2005-02

PRIMARY OUTCOMES:
Medication adherence based on pill counts

SECONDARY OUTCOMES:
Medication management ability

CONTACTS AND LOCATIONS:
Overall Officials: Sarah I Pratt, PhD, Principal Investigator — Assistant Professor in Psychiatry, Dartmouth Medical School
Locations (1):
- Community Council of Nashua, Nashua, New Hampshire, United States